CLINICAL TRIAL: NCT01388985
Title: Simplifying the Rabies Pre-exposure Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Military Hospital, Brussels (Unknown); Sciensano (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITMC0211; 2011-001612-62 (EudraCT Number)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Rabies
Keywords: Rabies; Vaccination; Boostability
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard vaccination schedule (Active Comparator): One injection will be given on three different days (day 0, day 7 and day 21 or 28)
  Interventions: Biological: Human Diploid Cell Vaccine (HDCV) rabies vaccine
- Accelerated vaccination schedule (Experimental): Two injections will be given on the same day (day 0 and day 7): one on each forearm.
  Interventions: Biological: Human Diploid Cell Vaccine (HDCV) rabies vaccine

INTERVENTIONS:
Biological: Human Diploid Cell Vaccine (HDCV) rabies vaccine — Human Diploid Cell Vaccine (HDCV) rabies Merieux 1 ml vaccine for rabies, provided by Sanofi-Pasteur, administered zvia ID route at two sites

SUMMARY:
Rabies is a viral zoonosis that causes an encephalitis, almost invariably fatal. It is widely distributed across the globe: the World Health Organization (WHO) estimates that about 2,4 billion people live in endemic areas for canine rabies. Vaccination of domestic animals is limited to industrialized and middle-income countries.

The development of clinical rabies can be prevented through timely immunization after exposure: however, preventive vaccination simplifies the post-exposure procedure considerably, as immunoglobulins are no longer needed and less vaccine administrations are scheduled. Pre-exposure prophylaxis consists of an intramuscular (IM)of intradermal (ID) dose given on days 0, 7 and 21 or 28. The development of immunological memory after this vaccination is critical for the establishment of long lasting immunity. Subjects receiving a booster dose 1 year after pre-exposure prophylaxis segregate themselves into 'good' and 'poor' responders; the former may not need further boosters for 10 years, whereas the latter may need more frequent boosters.

Until recently, guidelines in travel medicine recommended pre-exposure vaccination only for some risk groups. Since recent studies have shown the effectiveness of the ID vaccination, the policies are changing towards pre-exposure vaccination for a larger population, including travelers to endemic regions, where immunoglobulins and vaccine are often not readily available.

Based on the above, the investigators must stress the concept of "boostability" after a risk exposure. However, the current pre-exposure vaccination scheme could be improved: a schedule of 1 week would be less time consuming, would improve compliance and give less interference with other prophylaxis measures, e.g. mefloquine. Two small studies suggest that a schedule of 1 week interval is as effective and immunogenic as the standard one.

The investigators will investigate whether the accelerated schedule is as effective as the classical schedule, by carrying out a randomized, non-inferiority study.

DETAILED DESCRIPTION:
Rabies is a viral infection that affects the central nervous system and causes an encephalitis which is almost invariably fatal. Being a zoonosis, the infection usually occurs following a transdermal bite or scratch by an infected animal, but contamination may also occur when infectious material, usually saliva, comes into direct contact with the victim's mucosa or with fresh skin wounds. Human-to-human transmission is extremely uncommon.

Rabies is widely distributed across the globe: the World Health Organization (WHO) estimates that 87 countries with a total population of about 2,4 billion people are afflicted with endemic canine rabies, and the inclusion of all species poses a potential threat to >3.3 billion people. The number of rabid wild animals that die without being detected is however estimated to be more than 90% of the total, so identified infections represent only a small fraction of wild animal rabies cases. Vaccination of domestic animals is limited to industrialized nations, the most urbanized areas of Latin America and some Asian countries such as Thailand.

The development of clinical rabies can be prevented through timely immunization after exposure to the infecting agent: preventive vaccination alone implies no complete protection, but it simplifies the post-exposure procedure considerably, as immunoglobulins are no longer needed and less vaccine administrations are scheduled. Pre-exposure prophylaxis consists of an intramuscular (IM)of intradermal (ID) dose given on days 0, 7 and 21 or 28. The development of immunological memory after this vaccination is therefore critical for the establishment of long lasting immunity against rabies in humans. If a booster dose is given 1 year after pre-exposure prophylaxis, subjects segregate themselves into 'good' and 'poor' responders; the former group, who represent 75% of subjects, may not need further booster vaccination for 10 years, whereas the latter may need more frequent boosters.

Until recently, guidelines in travel medicine recommended the pre-exposure vaccination only to the classic risk groups. Since recent studies have shown the effectiveness of the ID vaccination, the policies are changing towards the recommendation of pre-exposure vaccination for a larger population, including all travelers to endemic regions, where rabies immunoglobulins and vaccine are often not readily available. The ID pre-exposure vaccination, which is more cost-effective, could also become an affordable alternative to protect the local population in high endemic regions.

Based on all the above, the investigators must stress the concept of "boostability" after a risk exposure: the main target of travel medicine today is to get a sufficient serological response on day 7 after a risk in prevaccinated persons (accelerated immune response through memory cells) and after two post-exposure vaccinations (day 0 and 3). It should also be noted that a schedule of 1 week would be preferable to the current schedule, because it would be less time consuming, would improve compliance and gives less interference with the intake of other prophylaxis measures, e.g. mefloquine. Two recent but small studies from Thailand suggest that an accelerated schedule of three intradermal injections within 1 week interval is as effective and immunogenic as administered within 4 weeks.

Therefore, this randomized, non-inferiority study will investigate whether the accelerated schedule is as effective as the classical schedule. The investigators will also increase the number of sites of injection, from one to two, to stimulate several different groups of lymph nodes on the same time to initiate more antibody production.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide written consent
* Seronegative for rabies
* Belgian soldiers who are deployable and visit the Travel clinic in Brussels during their preparation phase before deployment OR military students at the schools of Belgian Defense are eligible in preparation of an overseas exercise or during the scheduled vaccination program at the end of their studies
* Prepared to follow the study schedule

Exclusion Criteria:

* Subjects who have had rabies vaccination (complete or incomplete) in the past due to post-exposure prophylaxis.
* Subjects with a known allergy to one of the components of the vaccine.
* Immune depressed persons or intake of immunodepressant medication.
* Subjects who take mefloquine
* Planned deployment to overseas areas within 35 days.

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Soentjens, MD, Principal Investigator — ITM and Military Hospital
Locations (1):
- Military Hospital, Brussels, Belgium

REFERENCES:
- [Result] Soentjens P, Andries P, Aerssens A, Tsoumanis A, Ravinetto R, Heuninckx W, van Loen H, Brochier B, Van Gucht S, Van Damme P, Van Herrewege Y, Bottieau E. Preexposure Intradermal Rabies Vaccination: A Noninferiority Trial in Healthy Adults on Shortening the Vaccination Schedule From 28 to 7 Days. Clin Infect Dis. 2019 Feb 1;68(4):607-614. doi: 10.1093/cid/ciy513. PMID 29939243
- See also: EudraCT entry for the trial 2011-001612-62 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-001612-62/BE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants (1 in each group) signed the ICF and were randomized, but withdrew their consent before the first vaccination. They are not included in any of the analyses.
Period: Overall Study
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Started | 249 (1 participant (from the 250 enrolled) did not receive any vaccination because of consent withdrawal.) | 249 (1 participant (from the 250 enrolled) did not receive any vaccination because of consent withdrawal.)
Primary Vaccination Period | 231 | 238
Completed | 200 (From those 200, 15 were excluded from the per protocol analysis.) | 211 (From those 200, 28 were excluded from the per protocol analysis.)
Not Completed | 49 | 38
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 30 | 30
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Subject unavailable | 1 | 1
Not completed — Other (no reason) | 0 | 1
Not completed — Error of nurse | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule | Total
Number analyzed (Participants) | 249 | 249 | 498
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [24 to 35] | 28 [23 to 34] | 29 [23 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 237 | 241 | 478
Serology at baseline [Count of Participants; unit: Participants]
  0.5 IU/mL or less | 245 | 248 | 493
  more than 0.5 IU/mL | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Boostability of the Rabies Antibodies After Booster Vaccination
Description: The primary endpoint is the number of particpants with a boostability of the rabies antibodies on day 7 after booster vaccination, carried out at years 1 to 3 after initial vaccination. A rabies serology value of more than 0,5 IU/ml (international unit/milliliter) on day 7 after booster vaccination is considered to be protective. Subjects showing this serology value at day 7 are considered to be boostable.
Time Frame: Day 7 after booster vaccination
Population: From the total number of participants that completed the study (200 in the standard vaccination schedule and 211 in het accelerated vaccination schedule), not all were included in het per protocol analysis. 15 participants were excluded from the standard vaccination schedule group and 28 were excluded from the accelerated schedule group.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Number analyzed (Participants) | 185 | 183
Participants | 185 | 183

2. Secondary Outcome: Number of Participants With a Rabies Serology More Than 0.5IU/ml After Primary Vaccination
Description: Number of participants that have a Rabies serology more than 0,5 IU/ml on day 35 after primary vaccination.
Time Frame: Day 35 after primary (initial) vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Number analyzed (Participants) | 231 | 238
Participants | 231 | 238

3. Secondary Outcome: Number of Particpants With a Rabies Serology More Than 10IU/ml After Primary and Booster Vaccination
Description: Number of participants that have a Rabies serology more than 10 IU/ml on day 35 after primary vaccination, and after booster vaccination.
Time Frame: Day 35 after primary (initial) vaccination, and after booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Number analyzed (Participants) | 231 | 238
Participants | 189 | 167

4. Secondary Outcome: Number of Particpants Experiencing Adverse Events
Description: Number of participants experiencing Adverse events within one week after initial and booster vaccinations
Time Frame: One week after initial and booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Number analyzed (Participants) | 249 | 249
Participants | 190 | 190

5. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events
Description: Number of participants experiencing a Serious adverse event within 28 days after initial and booster vaccinations
Time Frame: 28 days after initial and booster vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
Number analyzed (Participants) | 249 | 249
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are collected until 1 week after the vaccination. Serious adverse events (SAEs) are collected until 28 days after the vaccination.
Arm/Group | Standard Vaccination Schedule | Accelerated Vaccination Schedule
All-Cause Mortality (participants affected / at risk) | 0/249 | 1/249
Serious Adverse Events (participants affected / at risk) | 1/249 | 2/249
Other Adverse Events (participants affected / at risk) | 0/249 | 0/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Vaccination Schedule (N=249) | Accelerated Vaccination Schedule (N=249)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemianopia (Nervous system disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes